CLINICAL TRIAL: NCT06374654
Title: Randomized Controlled Trial of Home-based Versus Formal Physical Therapy for Treatment of New Onset Non-insertional Achilles Tendinopathy
Brief Title: RCT of Home-based vs Formal Physical Therapy for Treatment of New Onset Non-insertional Achilles Tendinopathy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Chiodo, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P003272
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Protocol (Experimental)
  Interventions: Other: Home-based Exercise Protocol
- Formal Physical Therapy Protocol (Experimental)
  Interventions: Other: Formal Physical Therapy

INTERVENTIONS:
Other: Home-based Exercise Protocol — The home-based eccentric exercise protocol is a do-as-tolerated variation on the protocol described by Alfredson et al. in 1998. The protocol includes doing a series of heel raises, twice daily. No equipment is necessary. Patients will be given handouts and video links that depict and describe the exercises and their prescribed frequency.
  Arms: Home-based Protocol
Other: Formal Physical Therapy — Patients will be given a prescription for physical therapy consisting of 1-2 sessions per week for 6 weeks, with a renewal for another 6 weeks to be executed at the physical therapists' discretion. If an in-person visit is necessary for the renewal, or is requested by the physical therapist, the patient will be seen again in the office. Each patient will be given a release form to provide to his or her physical therapist. The release form will request a written record of all the treatment methods used by the physical therapist. Physical therapists who participate in the care of patients in this study will treat each patient using any and all methods that their professional experience deems clinically necessary.
  Arms: Formal Physical Therapy Protocol

SUMMARY:
The goal of this prospective randomized controlled trial is to compare the effectiveness of a home-based exercise protocol to formal physical therapy in patients who have been diagnosed with Achilles tendinopathy. The null hypothesis is that there will be no difference in the treatment outcomes between patients with Achilles tendinopathy who participate in a home-based program versus patients with Achilles tendinopathy who undergo formal physical therapy. Participants will be randomized to a 12-week home-based or formal physical therapy protocol and asked to complete brief outcomes surveys at their initial visit, and at 6 weeks, 12 weeks, 6 months, and 1 year after their initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age
* Must have a new diagnosis of Achilles tendinopathy that has presented with pain, thickening and tenderness at the mid substance of the Achilles tendon
* Symptoms present for at least 6 weeks

Exclusion Criteria:

* Patients with insertional Achilles pain or tenderness or concomitant plantar foot pain
* Patients who have had prior treatment with home eccentric stretching or physical therapy
* Patients who have prior diagnosis and treatment for Achilles tendinopathy
* Patients with history of injection (corticosteroid or sclerosing agents) to the Achilles tendon
* Patients with inflammatory arthritis
* Recent fluoroquinolone antibiotics (these agents are known to alter Achilles tendon physiology)
* Patients who have had prior foot or ankle surgery
* Individuals that do not speak English
* Bilateral disease
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2027-07-03 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment self-administered Achilles questionnaire (VISA-A) | Initial presentation, 6 weeks, 12 weeks, 6 months, and one year from the start of treatment
  Achilles tendon-specific questionnaire that asks about patient pain, functional status, and activity level.

SECONDARY OUTCOMES:
PROMIS Pain Interference (4a) | Initial presentation, 6 weeks, 12 weeks, 6 months, and one year from the start of treatment
PROMIS Pain Intensity (3a) | Initial presentation, 6 weeks, 12 weeks, 6 months, and one year from the start of treatment
PROMIS Depression (4a) | Initial presentation, 6 weeks, 12 weeks, 6 months, and one year from the start of treatment
Patient Acceptable Symptom State Questionnaire | Initial presentation, 6 weeks, 12 weeks, 6 months, and one year from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Chiodo, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No